CLINICAL TRIAL: NCT04470687
Title: Innovative Applications of Ultrafast Ultrasound Imaging in Peripheral Vascular Pathology: Evaluation of Carotid Plaque Vulnerability by Quantification of Neovascularization
Brief Title: Ultrafast Ultrasound Imaging Assesment of Carotid Plaque Neovascularization
Acronym: ULTRA-VASC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP180482; 2019-A03331-56 (Other: ANSM)
Record Dates: First submitted 2020-07-09; First posted 2020-07-14 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Carotid Stenosis; Carotid Artery Diseases; Carotid Atherosclerosis; Carotid Artery Plaque; Atheroma; Carotid Artery
Keywords: Carotid Stenosis; Endarterectomy, Carotid; Carotid Arteries; Carotid Artery, Internal; Stroke; Ultrasonography; Ultrasonography, Doppler; diagnostic imaging; Prognosis; Contrast Media
MeSH Terms: conditions — Carotid Stenosis; Carotid Artery Diseases; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Carotid plaque or stenosis ultrasound enhanced UF assesment (Experimental): symptomatic or asymptomatic patients with atheromatous carotid stenosis scheduled for carotid endarterectomy
  Interventions: Device: contrast enhanced ultrafast ultrasound imaging

INTERVENTIONS:
Device: contrast enhanced ultrafast ultrasound imaging — Ultrasound contrast medium: SonoVue 8µL/mL (Bracco International BV) Ultrasound scanner: Aixplorer® device marketed by SuperSonic Imagine©, CE Doppler UltraFast™Doppler, contrast ultrasound (CEUS), color Doppler and ultra-sensitive energy Doppler, high-performance directional energy Doppler, Elastography ShearWave™ UF-Doppler (UltraFast-Doppler) and microbubble injection (SonoVue) Apparatus for performing the UF Doppler sequence: Aixplorer, manufacturer : Supersonic Imagine, Aix-en-Provence, France, CE Marking.
  3D RCA dedicated vascular probe with dedicated Doppler sequences

SUMMARY:
Stroke is the second leading cause of death in the Western world and the leading cause of major lifelong disability. About 15% of strokes are secondary to thrombosis or embolization of an unstable atheromatous carotid plaque. In these symptomatic patients, the degree of carotid stenosis is correlated with the risk of early recurrence. Patients with stenosis over 70% are therefore offered an endarterectomy, an operation to remove carotid plaque, to prevent future strokes[1]. In asymptomatic patients, the degree of stenosis is a limited predictor, and better risk stratification is required to assess the degree of plaque vulnerability and stroke risk of the patient. The therapeutic decision towards endarterectomy in addition to drug therapy is debated because of a variable and dependent benefit/risk balance for each patient. A number of imaging parameters have been studied: ulceration, heterogeneity, vascularization of the plaque for example, but their place is not well defined [2].

The usual evaluation of carotid stenosis is by conventional Doppler ultrasound with calculation of the degree of stenosis according to the NASCET criteria.

For symptomatic stenoses the intervention is recommended when above 70% and is discussed from 50% to 70% of NASCET stenosis degree.

For asymptomatic stenoses, the procedure is discussed when above 60% taking into account the patient's life expectancy, the risk of the surgery and the unstable nature of the plaque [2].

Destabilization of the carotid plaque is partially induced by inflammation associated with neo-vascularization. The detection of these new vessels by conventional contrast ultrasound has already shown a distinction between stable and unstable plaques, by the presence or absence of microbubbles in the plaque. However, this assessment is not very precise and only the most vascularized plaques can be detected. Ultrafast ultrasound Imaging is a new ultrasonic Imaging modality that allows detecting low speed flows, a tiny vascular structure within the vessel wall.

RESEARCH HYPOTHESIS Plaques neo-vascularization would be more precisely detected and characterized by ultrafast imaging coupled with microbubble injection than conventional ultrasound imaging.

A better assessment of plaque instability could improve the selection of patients for carotid endarterectomy and increase the benefit/risk ratio of this preventive surgery.

DETAILED DESCRIPTION:
see above

ELIGIBILITY:
Inclusion Criteria:

* The patient is over 18
* The patient is scheduled for carotid endarterectomy within 30 days at most
* The patient has a social security system

Exclusion Criteria:

* Non-atheromatous carotid stenosis (radiation)
* Contraindication of the use of SonoVue ultrasound contrast media. Hypersensitivity to the active ingredient or any of the following excipients: Macrogol 4000; Distearoylphosphatidylcholine; Dipalmitoylphosphatidylglycerol sodium; Palmitic acid.
* The patient has any of the following conditions: right-left shunt, severe pulmonary hypertension (pulmonary blood pressure > 90 mm Hg), uncontrolled systemic hypertension and respiratory distress syndrome.
* Lack of social security coverage, patient under justice
* Allergy to ultrasound gel
* Pregnancy. (As a precautionary measure, it is best to avoid using SonoVue during pregnancy according to SPC)
* Patient under guardianship or curatorship or under the protection of justice.
* Patient unable or unwilling to give written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Neovascularization of the carotid plaque | end of inclusions
  Correlation BETWEEN the average signal strength of the carotid plaque analyzed after injection of ultrasound contrast medium by three-dimensional probe with UF-Doppler AND the number of neovessels determined by histological analysis of the carotid plaque (number of neovessels per section) studied.

SECONDARY OUTCOMES:
Plaque stable or unstable | end of inclusions
  analyzed after injection of ultrasound contrast medium by three-dimensional probe with UF-Doppler AND the plaque stability according to Oxford criteria
Plaque symptomatic or not | end of inclusions
  Comparison BETWEEN the average signal strength of the carotid plaque analyzed after injection of ultrasound contrast medium by three-dimensional probe with UF-Doppler AND the symptomatic or asymptomatic status for stroke of the patient

CONTACTS AND LOCATIONS:
Overall Officials: Tristan MIRAULT, MD, PhD, Principal Investigator — Hopital europeen Georges-Pompidou
Locations (1):
- Hopital europeen Georges-Pompidou, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared
Supporting Information: Study Protocol, ICF
Time Frame: Data could be available one year after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on scientific project and scientific involvement of the PI team.
  Teams wishing obtain IPD must meet the sponsor and IP team to present scientifics (and potentially commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractualization.